CLINICAL TRIAL: NCT02177058
Title: Implementing Interventions to Reduce Hospitalizations of Nursing Home Residents
Brief Title: Reducing Hospitalizations of Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 304897; 5R01NR012936-02 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-03

CONDITIONS: Unnecessary Hospitalizations of Nursing Home Residents
Keywords: Nursing homes; Hospitalizations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immediate INTERACT implementation (Experimental): INTERACT Quality improvement program training and implementation between APR 2013 and MAR 2014
  Interventions: Other: INTERACT Quality improvement program
- Delayed intervention with reporting (Active Comparator): Quarterly surveys/data reporting between APR 2013 and MAR 2014. They receive INTERACT training starting on MAR 2014.
  Interventions: Other: Quarterly surveys/data reporting
- Delayed intervention not reporting (No Intervention): No data collected from these nursing homes for one year since baseline. They receive INTERACT training starting on MAR 2014.

INTERVENTIONS:
Other: INTERACT Quality improvement program — INTERACT training and implementation between APR 2013 and MAR 2014
  Arms: Immediate INTERACT implementation
Other: Quarterly surveys/data reporting — The nursing homes are asked to complete quarterly surveys between APR 2013 to MAR 2014
  Arms: Delayed intervention with reporting

SUMMARY:
This project directly addresses the national imperative for innovative strategies to improve care for Medicare beneficiaries and reduce health care costs. The overall objective of the proposed project is to improve the care of older individuals who reside in nursing homes (NHs), and at the same time reduce unnecessary Medicare expenditures. This goal will be accomplished by testing a quality improvement program designed to reduce the number of avoidable hospitalizations of NH residents in a randomized controlled trial.

The primary hypotheses to be tested are:

Hypothesis1: Interventions to Reduce Acute Care Transfers (INTERACT) implementation NHs will have a greater reduction in hospitalization rate than the control and monitoring only NHs during the 12-month implementation compared to a 12-month baseline period.

Hypothesis 2: Reductions in Medicare expenditures for hospitalizations in the INTERACT implementation NHs will be greater than the estimated costs of implementing the intervention.

Hypothesis 3: The effects of INTERACT on hospitalization rates will be greater among patients on the Medicare skilled benefit for post-acute care, than for long-stay patients.

Hypothesis 4: The effects of INTERACT on hospitalization rates will be greatest among those NHs with higher vs. lower intensity (fidelity) of implementing the program.

Hypothesis 5: There will be a greater reduction in measures of hospitalizations for conditions defined as "potentially preventable" than for other transfers and hospitalizations.

Hypothesis 6: Implementation of INTERACT will not be associated with worsening of relevant quality measures in the participating NHs.

DETAILED DESCRIPTION:
Hospitalizations of Nursing Home (NH) residents are frequent and associated with numerous complications and increased health care costs. Previous research suggests that as many as two-thirds of such hospitalizations may be avoidable. Anticipated changes in Medicare reimbursement will reduce financial incentives that favor hospitalization, but could result in reduced care quality if NH staff does not have the training and clinical tools to manage residents in the NH when acute changes occur. INTERACT (Interventions to Reduce Acute Care Transfers) is a quality improvement program that utilizes tools based on established clinical guidelines. The tools target three key strategies to reduce potentially avoidable hospitalizations: 1) preventing conditions from becoming severe enough to require acute hospital care; 2) managing selected acute conditions in the NH; and 3) improving advance care planning for residents among whom a palliative or comfort care plan, rather than acute hospitalization, may be appropriate. Preliminary research involving 30 NHs demonstrated a 17% reduction in hospitalizations compared to the same six-month period in the previous year. The cost of the intervention was $7,700; projected savings to Medicare of reduced hospital admissions from a 100-bed NH were $125,000/year. While these results are promising, the effectiveness of INTERACT in reducing hospitalizations remains to be tested in a controlled trial. The proposed project will therefore involve an interdisciplinary team of experienced NH researchers in conducting a randomized controlled trial to test the implementation of the INTERACT program. NHs randomized to the INTERACT intervention will participate in 3-months of training, and receive support during the 12-month implementation period by an experienced nurse practitioner through regular multi-NH conference calls, monthly individual calls, and as-needed telephonic or email communication. The effects of implementing the INTERACT intervention on hospitalization rates will be compared to a randomly assigned group of usual care control NHs and a group that will self-monitor hospitalization rates only. The hypotheses to be tested are:

1) INTERACT implementation NHs will have a greater reduction in hospitalization rates than the control and monitoring only NHs during the 12-month implementation compared to a 12-month baseline period; and 2) reductions in Medicare expenditures for hospitalizations in the INTERACT intervention NHs will exceed the estimated costs of implementing the intervention.

The specific aims of this project are to:

1. Determine the effectiveness of implementing the INTERACT quality improvement program in reducing hospitalization rates.
2. Calculate the differences in Medicare expenditures for hospitalizations between NHs implementing INTERACT, the usual care control group, and NHs in the monitoring hospitalization rates only group.

ELIGIBILITY:
Inclusion Criteria:

* > 40 Beds
* MD, NP or PA available on-site at least 1/week
* Capable of Starting intravenous fluids
* Capable of Providing respiratory treatments
* Capable of Assessing oxygenation status by pulse oximetry
* < 4 hrs turnaround time for STAT medications ("stat" is an abbreviation of the Latin word statim, meaning "immediately, without delay")
* < 8 hrs. turnaround time for STAT laboratory tests
* < 8 hrs. turnaround time for STAT X-rays
* Computers available for online staff training
* Strong support for participation from the facility administrator, director of nursing, and medical director, as well as corporate leadership (for NHs that are part of a corporate chain), as evidenced by a signed agreement before enrollment
* > 10% 30-day readmission rates

Exclusion Criteria:

* Hospital based
* Having only private pay residents (no Medicare/Medicaid, no Medicare provider number).
* Participation in a project designed specifically to reduce acute care transfers or hospitalization rates (including federal demonstrations)
* Conducting more than one other major quality improvement or research project during the project period which would threaten their ability to fully participate in the trial.
* Specialize in Pediatrics (> 30 % of patients in NHs are pediatric)
* Specialize in HIV (> 30 % of patients in NHs are HIV)
* Specialize in Respiratory care with ventilator care (>30% of patients in NH are in this category)
* Robust INTERACT implementation and/or very low hospitalization rate
* Located in a country outside USA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Reductions in hospitalization | 1 year

SECONDARY OUTCOMES:
Reduction in hospitalization rates during high-risk periods and low-risk periods. | 30 days
  High Risk Periods: within 30-day of NH admission. Low risk period: ≥31 days after NH admission.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G Ouslander, MD, Principal Investigator — Florida Atlantic University; Ruth M Tappen, EdD RN FAAN, Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University, College of Medicine/College of Nursing, Boca Raton, Florida, United States

REFERENCES:
- [Derived] Tappen RM, Newman D, Huckfeldt P, Yang Z, Engstrom G, Wolf DG, Shutes J, Rojido C, Ouslander JG. Evaluation of Nursing Facility Resident Safety During Implementation of the INTERACT Quality Improvement Program. J Am Med Dir Assoc. 2018 Oct;19(10):907-913.e1. doi: 10.1016/j.jamda.2018.06.017. Epub 2018 Aug 11. PMID 30108035
- [Derived] Kane RL, Huckfeldt P, Tappen R, Engstrom G, Rojido C, Newman D, Yang Z, Ouslander JG. Effects of an Intervention to Reduce Hospitalizations From Nursing Homes: A Randomized Implementation Trial of the INTERACT Program. JAMA Intern Med. 2017 Sep 1;177(9):1257-1264. doi: 10.1001/jamainternmed.2017.2657. PMID 28672291
- [Derived] Ouslander JG, Naharci I, Engstrom G, Shutes J, Wolf DG, Rojido M, Tappen R, Newman D. Hospital Transfers of Skilled Nursing Facility (SNF) Patients Within 48 Hours and 30 Days After SNF Admission. J Am Med Dir Assoc. 2016 Sep 1;17(9):839-45. doi: 10.1016/j.jamda.2016.05.021. Epub 2016 Jun 24. PMID 27349621
- See also: Related Info — http://www.pathway-interact.com/